Using Motivating Reminiscence Technology to Encourage Physical Activity and Improve Balance and Mobility for Residents in Long Term Care.

Bruyere REB Number: M16-19-012

University of Ottawa REB Number: H-05-19-4462

Ottawa Health Science Network REB Number: 20190454-01H

ClinicalTrials.gov Identifier: NCT04043416



Project Protocol

May 2019

### 1. Project Team

### Elizabeth Bruyère Primary Investigator:

Dr. T Mark Campbell, MD Clinician Investigator Elizabeth Bruyère Hospital tcampbell@bruyere.org

### **Project Lead:**

Susan Zorz
Director of Resident Services
The Glebe Centre Inc.
SZorz@glebecentre.ca
Ph. 613.238.2727 X 323
Fx. 613.238.4759

### **Co-Investigators**

Becky MacLeod Recreation Therapist The Glebe Centre Inc 613-238-2727 bmacleod@glebecentre.ca

Suja Thomas Coordinator of Nursing Programs The Glebe Centre Inc sthomas@glebecentre.ca

Sean Dellaire Research Associate The Glebe Centre Inc

Kathryn L May, NP Nurse Practitioner The Ottawa Hospital Kmay@toh.ca

### **Study Administration Assistant:**

Katherine Reilly University of Ottawa 613-562-5800 x8238 kreilly@ohri.ca

### 2. Title

Using Motivating Reminiscence Technology to Encourage Physical Activity and Improve Balance and Mobility for Residents in Long Term Care.

### 3. Background

Physical activity has numerous benefits for physical well-being and function in the elderly<sup>2</sup>. Maintaining the functional independence of Long-Term Care (LTC) residents alleviates the everincreasing demands placed on front line staff. Physical activity also provides an opportunity for LTC residents to engage in valued activity<sup>3</sup>. However, many LTC residents rarely or never engage in regular physical activity due to numerous barriers such as lack of exercise equipment or related resources and lack of interest or motivation<sup>4</sup>. For these reasons, adults residing in LTC facilities have been shown to have drastically lower physical activity levels<sup>5</sup>. Those who do engage in regular physical activity maintain functioning and reduce negative health outcomes including but not limited to deconditioning, falls and cognitive decline<sup>1</sup>. For the positive effects of physical activity to last, it is essential that training becomes routine, meaning that easy access and proximity to training opportunities as well as the provision of engaging modalities is of great importance.

A stationary bicycle is a type of exercise equipment that resembles a bicycle without wheels and can engage a user in a similar way standard bicycling can. Stationary cycling is one example of a physical activity modality that provides opportunities for meaningful activity for LTC residents. Advantages of stationary cycling include limited space requirements, lower risk of harm or resources compared to activities such as swimming or walking outside with a population with dementia or mild cognitive impairment. Balance control has been shown to be less deteriorated for older individuals that engage in outdoor cycling activity<sup>7,8</sup> perhaps due to an observed improvement in muscle strength and power with parallel increases in walking speed and other functional abilities<sup>9</sup>. Cycling activity is also beneficial for maintaining cognitive performance across multiple domains for older institutionalized individuals<sup>6</sup>. One of the challenges associated with stationary physical activity however is that it may be perceived as dull or disengaging. Novel ways to engage older adults is therefore of great importance in order to maintain a regular fitness program.

Reminiscence is defined as inducing a vocal or silent recall of past activities, events, and experiences in the life of a person by using tangible prompts<sup>10</sup>, has been shown to be effective in improving cognitive functions while reducing depressive symptoms<sup>11</sup>. The ability to select specific virtual cycle trips according to the users' wishes and memories may increase reminiscence for that individual and, when coupled with a stationary cycling intervention, increase motivation for that physical activity.

The use of jDome BikeAround provides older adults in LTC an opportunity to engage in a motivating reminiscence activity that is coupled with physical activity that may have positive impact on maintaining physical and cognitive abilities thereby maintaining function and reducing fall risk.

### 4. Rationale

One of the biggest challenges faced in LTC is to offer meaningful activities to residents. The jDome BikeAround system provides an ideal opportunity to explore the impact of targeted, specific activity interventions for people who have significant cognitive issues and other chronic health conditions and disabilities. This specific system has never been examined within the literature or any small scale published studies of the benefit of the BikeAround system, highlighting the need to examine this system in a controlled study.

The BikeAround uses Google Street View, a stationary bike and a domed screen (Figure 1). Residents are seated in front of the screen; their destination is typed into the computer and when loaded the image appears on the screen. Using pedals on the bike they can propel themselves down the street, steer and change direction as they wish. Residents are able to visit familiar places anywhere in the world or travel to places they have always wanted to visit. Discussion of past activities, events and experiences will be aided by visited locations and conversations with cycle hosts (i.e. trained staff/volunteers). We will use a mixed methods approach to explore the feasibility and impact of our individualized, personalized structured programs.

The BikeAround system is an innovative program that encourages reminiscence, physical and cognitive stimulation and is a fun activity that promotes positive, interactive experience. This project aims to identify the physical benefits of using a jDome BikeAround reminiscence physical activity program for LTC residents.



Figure 1: jDome BikeAround Set-up.

Image source: https://www.camanio.com/us/products/bikearound/

### 5. Objectives

- 1. Determine whether there are any effects on outcome measures of balance, mobility and fall risk reduction from the addition of jDome BikeAround
- 2. Determine whether reminiscence is facilitated through the observation of locations from jDome BikeAround.
- 3. Determine feasibility of integrating the technology into care on the units at the Glebe Centre.

### 6. Hypotheses

- 1. Residents will have an improvement in their balance, mobility, and fall risk as shown by the physical outcomes due to an enjoyable interaction with the jDome BikeAround that stimulates reminiscence and increased physical activity for residence at the Glebe Centre;
- 2. The reminiscence is facilitated through the observation of locations from the jDome BikeAround;
- 3. Integrating the jDome BikeAround technology into care at the Glebe Centre is feasible;

### 7. Outcomes

Primary Outcomes

- 1. Feasibility
  - a. The ability to enroll 30 participants from The Glebe Centre
  - b. Number of participants who completed the protocol
  - c. Number of adverse events
- 2. Physical Outcome Measures (Appendix A)
  - a. Tinetti Performance-Oriented Mobility Assessment (POMA) scale

### Secondary Outcomes

- 1. Participation (Appendix B)
  - a. Sessions attended

(Reasons for not attending scheduled sessions)

- b. Total number of sessions
- c. Total time per session
- d. Distance traveled
- e. Wong Baker Scale to evaluate satisfaction
- f. Resistance
- 2. Qualitative feedback/field notes (Appendix C)
- 3. Physical Outcomes
  - a. Knee Range of Motion
  - b. Two Minute Walk Test (TMWT)
- 4. Chart Data from the CIHI quarterly reports, RAI-MDS and Activity-PRO reporting mechanisms. (Appendix D)
  - a. Number of falls during previous year
  - b. Cognitive Performance Scale (CPS)
  - c. Revised Index of Social Engagement (RISE)

### 8. Methods

### 1. Study Design

This research project will use a cross-over pre-post study design (Appendix E) to collect mixed methods data for up to 30 participants. Each phase will last 6 weeks. A washout phase (phase 2) will allow the residents to also serve as their own comparison groups. The washout period is intended to allow activity levels to return to baseline between the two phases.

### 2. Study population, sample selection/consent process and sample size justification

The study population will consist of residents from the 254-bed Glebe Centre Residence (Ottawa, ON). Recruitment of the participants will commence with a notification going out through the Glebe Centre Newsletter. The small paragraph (Appendix F) will inform readers that a research project will be underway and may be appropriate for them/their resident. There will also be a poster put up in the main foyer to advertise the study (Appendix N). The poster was initially presented at the 2018 Regional Geriatric Annual General Meeting and will be repurposed as an advertisement tool. Contact information for the research team will be included if more information is required.

We will aim to recruit participants of varying age groups (though participants must be  $\geq 18$  years), sex/gender, and who are able to complete the outcome measures (Section 7, Outcomes).

### **Inclusion Criteria**:

- a. Scott fall risk of 2-17 (this is the current range used by the Glebe Centre, there have been 0 falls during transportation to the equipment and during each session of the BikeAround system)
- b. Sufficient visual abilities to observe images on the domed screen
- c. Able to comprehend and communicate in English.
- d. Adequate attentional capacity to remain focused on the pedalling task.
- e. Minimum height requirement of 5'2" or 157cm in order to successfully fit the BikeAround system's stationary bike.

We will exclude residents with the following, as determined by the Glebe Centre healthcare team:

- Physical limitations (as determined by the Glebe Centre healthcare/physiotherapy team) that prevent use of the jDome bike.
- Cognitive impairment (as determined by the Glebe Centre healthcare/physiotherapy team)
  - Inability to sustain attention
  - o Inability to follow one-step commands.
- Known behavioural abnormalities (e.g. overly aggressive behavior) that in the opinion of the clinical care team might impede any meaningful participation in the project
- Those who are in the opinion of attending physician or clinical team too unwell to participate in the project
- Fully unable to complete outcome measures indicated (Section 7, Outcomes)

Late exclusions may occur if the resident's condition declines after providing consent such that they then meet exclusion criteria.

Inclusion and exclusion criteria for participation will be made known to a member of the resident's primary circle of care who will inform potentially eligible residents of the opportunity to participate in the study. This staff member will ask if the resident would like to provide contact information to a member of the research team (who will not be a part of the primary circle of care) for the purpose of discussing study participation in more detail (see Recruitment Script for Staff; Appendix G). Agreement to discuss the project with a research team member will be documented on the patient's chart. In the event that the investigators are part of the resident's circle of care, they will neither be recruiting participants nor obtaining consent.

If the resident agrees to provide their name and room number, the member of the circle of care will forward the resident name and room number to the research assistant (RA) in a secure manner via password-protected voicemail and/or encrypted email. The RA will then visit the resident in-person (visit #1) on the unit to discuss the project (using Recruitment Script for RA; Appendix H) and obtain informed consent in-person (Appendix I). Potential participants and/or substitute decision-makers will be given an opportunity to read the consent form, ask questions and will be provided adequate time to make their decision.

Residents that are identified by the staff as being potential participants, but do not have the capacity to provide informed consent will not be excluded. If they are eligible but unable to provide informed consent (that is, they have a substitute decision-maker for their medical care), the substitute decision maker (SDM) will be contacted. The SDM on file will be contacted by a member of the resident's healthcare team and will be asked for verbal or written (via email) consent to provide contact information to the research team if they express interest in more information about their resident's participation in the study. A member of the research team will then call the SDM to obtain informed consent (Appendix J) for their resident. An option for the SDM to return their consent to participate in the research study either verbally or over email as it is possible that some will not be able to scan and send a signed consent form.

As per the Partnership of Consent Protocol<sup>12</sup>, after the SDM provides informed consent for the resident, assent is still required from the resident. If the resident provides no signs of dissent (shrieking, repetitive verbalizations, facial grimacing, hand wringing, or rocking movements), then the resident will be included in the study. However, if the resident shows signs of dissent, the behaviours will be verified with the LTC staff. If these signs are at baseline for that resident, it can be considered assent and the resident will be included. If the behaviours are not at baseline, the RA will wait 24 hours and try to approach the resident again. If the resident shows signs of dissent not at baseline for a second time, the resident will be excluded from participation in the study.

It is important that the patient also demonstrates assent for each jDome BikeAround session. Timing of each session will be optimized for each participant's daily schedule and activity performance. If the patient shows no signs of dissent before and during each jDome BikeAround session the session will continue. If the patient does show signs of dissent, or exhibits behaviour suggesting they are no longer willing to participate, the session will be ended. The patient will

be approached for another session 24 hours later, if the patient shows signs of dissent during the second attempt at a jDome BikeAround session that session will be halted and the patient will be withdrawn from the study.

### Sample Size

Sample size will be based upon our primary feasibility outcome. At the Glebe LTC, approximately 50 residents use the jDome BikeAround System annually. We estimate that over the course of the study timeframe that ~40% of these residents will be unavailable to participate. Thus, we expect to recruit 30 participants into the study. It should be noted that there are no other studies running at The Glebe Centre at the moment. Those that currently use the BikeAround system can be recruited into the study, but will undergo at least a 4-week washout period (no use of the system) prior to their initial participation in the study.

### 3. Methods and procedures for data collection and analysis

### ii. Data Collection

All participants will be assessed with the physical outcome measures (Section 7) prior to the commencement of the intervention (phase 1) as well as after each phase (total of 4 outcome measure time points, see Appendix E). Physical outcome measures will be done by a member of the physiotherapy team who will be blinded to the participants' current phase. Each measurement session is expected to take approximately 20 minutes and will include the POMA, 2MWT and knee ROM. Hard-copy versions of the all the data forms will not use resident identifiers but will instead use research team allocated study-specific identifiers that cannot be linked back to the participant (e.g. P01). All hard copies of study data will be kept in the physio team's locked office within a locked filing cabinet. All electronic and hard copies of study data will be destroyed and/or shredded 10 years after the culmination of the study. The masterlist that connects the study specific identifiers to the participants will be stored separately in a password-protected file on the Glebe's secure server.

Following the completion of pre-intervention outcome measures, the participants will be randomized into one of two possible groups Residents will either participate in the intervention during phase 1 or be delayed until phase 3. Due to the nature of the cross-over design, it is possible that participants will identify their group allocation (e.g. if their use of the jDome BikeAround System is delayed). This may result in performance bias, and is a limitation of our protocol. The physiotherapy team performing the outcome measures will be blinded to the group allocation, reducing the likelihood of detection bias. As per the standard of care all the patients will be participating in the 'fall prevention program' throughout all phases of the protocol. The standard fall prevention program involves reducing the incidence of residents' falls and mitigating risks of falls through a resident focused, team approach which ensures that a resident's environment and social, physical, cognitive and emotional strengths are supported. A more in-depth summary of the program can be found in Appendix L.

Data extraction of chart data will be completed by a research associate using a de-identified Microsoft Excel spreadsheet saved on the secure Glebe Centre server. A password-protected master list saved on the secure Glebe Centre server will contain resident identifying information and study identification codes and will be updated throughout the course of the study (Appendix K).

Personal health information extracted from the charts for the purposes of the study will include:

- a) Age
- b) Sex (Male, Female, or Other)
- c) Height
- d) Weight
- e) Medical diagnoses
- f) List of medications
- g) Cognitive Performance Scale score
- h) Revised Index of Social Engagement (RISE) score
- i) ActivityPro data
- ii. Analysis

### **Qualitative Analysis**

Qualitative field notes will be de-identified and imported into NVivo 11, a qualitative software program. Transcripts and field notes will be reviewed and coded using an iterative content analysis approach. Themes and sub-themes across transcripts will be identified using NVivo.

### **Quantitative Analysis**

We will determine the success of the primary outcome of feasibility as follows: 1) We are able to recruit 30 participants into the study; 2) Less than 15% of participants will be unable to complete the study; 3) There are no serious adverse events, defined as (i) major change in medical condition, injury, or intractable dizziness ± nausea related to the use of the jDome BikeAround System, (ii) severe emotional distress necessitating cessation of use of the jDome BikeAround System, (iii) falls either during transport to and from, or while using the jDome BikeAround System.

Regarding the primary physical outcome, POMA, we do not have data upon which to perform a power analysis for this part of the study, thus we are unable to set specific thresholds for success based on our available sample size.

All quantitative data (e.g. physical outcomes, participation data) will be analyzed using SPSS software with an  $\alpha$  of 0.05. Data will be analyzed to determine normality and appropriate statistical tests will be used to determine intergroup differences. Continuous data will be evaluated using methods such as student's t-test, categorical data will be evaluated using chi-squared.

### **Analysis Location**

All de-identified data will be entered into excel databases. This data will be transported on an encrypted external hard drive to the University of Ottawa where it will be stored on the Campbell Laboratory server space for data analysis. The data being transferred will not include the master list that connects study identifiers to individual participants and the data will only be transferred after the study intervention is complete.

### 4. Intervention details

In collaboration with the healthcare team and the residents, cycling sessions will be scheduled to provide consistency for the residents. A goal of 3 sessions every week will be attempted, this is the number of sessions attempted during regular implementation at the Glebe Centre. Each session will be facilitated by a "Cycle Host". A cycle host is either a trained staff or volunteer at the Glebe Centre. All Cycle Hosts will be required to undergo a 1-hour training session to ensure consistency between hosts and safety of the residents as well as how to assess whether the patients are giving ongoing consent. They may also provide basic technical support. The RA will also work closely with the participant's circle of care to ensure that the patients continue to meet the inclusion criteria. The cycle host will find the resident and bring them to the BikeAround and escort them back to their room following the session. The length of each BikeAround session will be at the participant's discretion provided the cycle host (research associate/volunteer) deem it safe and it does not exceed 30 minutes in one session, a common participation duration for current Glebe LTC resident users.

The jDome BikeAround sessions involve the use of Google Street View, a stationary bike and a domed screen. Residents are seated comfortably in front of the screen; their destination is typed into the computer and when loaded the image appears on the screen. Using pedals on the bike they can propel themselves down the street, steer and change direction as they wish. Residents are able to visit familiar places of their choosing anywhere in the world or travel to places they have always wanted to visit. As long as it has been mapped by Google, it can be displayed on the domed screen. Google StreetView covers 39 countries and approximately 3000 cities. Each session the participants have the option to pick their location, or the cyclehost can pick from preselected locations given by families and/or SDMs of the participants.

### 9. Risks/Benefits

We predict that there are minimal risks involved in participation in this study, though there is a chance of emotional distress being triggered by reminiscences. In the event that a participant begins to show signs of severe emotional distress, participation will be stopped immediately at the participant's request, and clinical chaplains and social workers will be available on the unit and contacted as soon as possible. The resident's attending physician and nurse will also be notified of any emotional distress caused as a result of this project.

It should be noted that with the regular use of the BikeAround system at the Glebe Centre over the last 12 months. During this time period there have been hundreds of sessions with over 50 residents have used the equipment multiple times per week. Only where 3 residents experienced adverse events during one of their sessions. All of them being that the resident felt dizzy during the session due to the speed the bike was appearing to be going on the screen. These adverse events have been resolved by changing the parameters of the jDome BikeAround session, where the speed of the video aspect is slowed and not dependent on the speed the participant is pedaling. The highest resident's Scott Fall Risk that has used the system in the past was 17, and there were no serious adverse events experienced.

Benefits to the residents may be limited to interaction with the jDome BikeAround with possible improvements to their balance and mobility. Increased social and psychological well-being may be possible as enjoyable reminiscence through videos/pictures have been shown to be a positive experience for individuals with dementia.

### 10. Timelines

**September – December 2018** Protocol and REB application development and submission

**December 2018 – February 2019** REB approval / liaison with REB to obtain approval

February - July 2019 Participant recruitment and data collection

**July – September 2019** Data analysis, synthesis of final report of findings

### 11. Potential Conflicts of Interest

The Glebe Centre is receiving financial payment from the Canadian Aging and Brain Health Innovation (CABHI) to cover the cost of conducting this study.

### 12. Contingency Planning

In the event of an epidemic, pandemic, or similar emergency situation where the research staff would not have access to the research participants the participants would not participate in the BikeAround system during that period. This would not affect the overall health of the participants since they will still be receiving the standard of care provided by staff at The Glebe Centre and would be cared for following the Glebe Centre's standard operating procedures during emergency situations.

### 13. Budget

See Appendix K

### 14. Publication and Dissemination of Results

The results of this study will be published in a peer-review journal and presented at national and international conferences. A summary of the results will also be included in the Glebe Centre's Newsletter, which will also be disseminated directly to the study participants.

### 15. Troubleshooting

Although highly unlikely due to the large available participant pool to draw from, in the case that not enough participants are available for recruitment, the information gathered will still be of use as this is the first research project on the use of the jDome BikeAround system for residents in long term care. The smaller sample size will impact the strength of significance but still provide a platform for future research.

### 16. References

- 1. Lautenschlager NT, Cox K, Kurz AF. Physical Activity and Mild Cognitive Impairment and Alzheimer's Disease. Curr. Neurol. Neurosci. Rep. [Internet]. 2010;10:352–8. Available from: http://link.springer.com/10.1007/s11910-010-0121-7
- 2. Vogel T, Brechat P-H, Leprêtre P-M, Kaltenbach G, Berthel M, Lonsdorfer J. Health

- benefits of physical activity in older patients: a review. Int. J. Clin. Pract. [Internet]. 2009;63:303–20. Available from: http://doi.wiley.com/10.1111/j.1742-1241.2008.01957.x
- 3. Menne HL, Johnson JD, Whitlatch CJ, Schwartz SM. Activity Preferences of Persons With Dementia. Act. Adapt. Aging. 2012;36:195–213.
- 4. Benjamin K, Edwards N, Ploeg J, Legault F. Barriers to physical activity and restorative care for residents in long-term care: a review of the literature. J. Aging Phys. Act. [Internet]. 2014;22:154–65. Available from: http://osearch.ebscohost.com.library.ucc.ie/login.aspx?direct=true&db=rzh&AN=107880169&sit e=ehost-live%5Cn10.1123/JAPA:2012-0139%5Cnhttp://osearch.ebscohost.com.library.ucc.ie/login.aspx?direct=true&db=ssf&AN=93710219&site=ehost-live
- 5. de Hollander EL, Proper KI. Physical activity levels of adults with various physical disabilities. Prev. Med. reports [Internet]. 2018;10:370–6. Available from: https://doi.org/10.1016/j.pmedr.2018.04.017
- 6. Varela S, Cancela JM, Seijo-Martinez M, Ayán C. Self-Paced Cycling Improves Cognition on Institutionalized Older Adults Without Known Cognitive Impairment: A 15-Month Randomized Controlled Trial. J. Aging Phys. Act. [Internet]. 2018;26:614–23. Available from: https://journals.humankinetics.com/doi/10.1123/japa.2017-0135
- 7. Batcir S, Melzer I. Daily Bicycling in Older Adults May be Effective to Reduce Fall Risks—A Case-Control Study. J. Aging Phys. Act. [Internet]. 2018;26:570–6. Available from: http://journals.humankinetics.com/doi/10.1123/japa.2017-0263
- 8. Harvey S, Rissel C, Pijnappels M. Associations Between Bicycling and Reduced Fall-Related Physical Performance in Older Adults. J. Aging Phys. Act. [Internet]. 2018;26:514–9. Available from: http://journals.humankinetics.com/doi/10.1123/japa.2017-0243
- 9. Macaluso A, Young A, Gibb KS, Rowe DA, De Vito G. Cycling as a novel approach to resistance training increases muscle strength, power, and selected functional abilities in healthy older women. J. Appl. Physiol. [Internet]. 2003;95:2544–53. Available from: http://www.ncbi.nlm.nih.gov/pubmed/12937026
- 10. Huang H, Chen Y, Chen P. Reminiscence Therapy Improves Cognitive Functions and Reduces Depressive Symptoms in Elderly People With Dementia: A Meta-Analysis of Randomized Controlled Trials. J. Am. Med. Dir. Assoc. [Internet]. 2015;16:1087–94. Available from: http://dx.doi.org/10.1016/j.jamda.2015.07.010
- 11. Karssemeijer EGA, Aaronson JA, Bossers WJ, Smits T, Olde Rikkert MGM, Kessels RPC. Positive effects of combined cognitive and physical exercise training on cognitive function in older adults with mild cognitive impairment or dementia: A meta-analysis. Ageing Res Rev. [Internet]. 2017; 40:75-83. Available from: <a href="https://www.sciencedirect.com/science/article/pii/S1568163717301149?via%3Dihub">https://www.sciencedirect.com/science/article/pii/S1568163717301149?via%3Dihub</a>
- 12. Batchelor-Aselage M, Amella E, Zapka J, Mueller M, Beck C. Research with dementia patients in the nursing home setting: a protocol for informed consent and assent. IRB [Internet]. 2014;36:14–20. Available from: http://www.ncbi.nlm.nih.gov/pubmed/24783377

### 17. Appendices

Appendix A – Physical Outcome Measures (Primary and Secondary)

Appendix B – Participation Log

Appendix C – Field Note Page

Appendix D – Medical Chart Data Outcome Extraction Sheet

Appendix E – Cross-over Study Design Diagram

Appendix F – Newsletter Paragraph

Appendix G – Recruitment Script for Staff

Appendix H – Recruitment Script For RA

Appendix I – Participant Consent Form

Appendix J – SDM Participant Consent Form

Appendix K – Master List Sheet

Appendix L – CABHI Budget

Appendix M – Summary of Fall Prevention Program at The Glebe Centre

Appendix N – Poster for presentation in main fover

### **Appendix A:** Physical Outcomes

### 17.1.1 <u>Demographic sheet</u>

| <u>Item</u> | <u>Value</u> |
|----------------------------------|--------------|
| Participant Number | |
| Gender | |
| D.O.B<br>(dd-mm-yyyy) | |
| Height (m) | |
| Weight (kg) | |
| Scott Fall Risk | |
| Number of falls in the past year | |
| Gait Aid Used (Y/N) | |

### 17.1.2 The Tinetti Test (Performance Oriented Mobility Assessment (POMA))

### DESCRIPTION

The Tinetti Assessment Tool is a simple, easily administered test that measures a resident's gait and balance. The test is scored on the resident's ability to perform specific tasks.

### TIME TO COMPLETE

10 to 15 minutes

### **SCORING**

Scoring of the Tinetti Assessment Tool is done on a three-point ordinal scale with a range of 0 to 2. A score of 0 represents the most impairment, while a score of 2 represents independence. The individual scores are then combined to form three measures; an overall gait assessment score, and overall balance assessment score, ad a combined gait and balance score.

### INTERPRETATION

The maximum score for the gait component is 12 points. The maximum score for the balance component is 16 points. The maximum total score is 28 points. IN general, residents who score below 19 are at a high risk for falls. Residents who score in the range of 19 - 24 points indicate that the resident has a risk for falls.

### RELIABILITY

Interrater reliability was measured in a study of 15 residents by having a physician and a nurse test the residents at the same time. Agreement was found on over 85% of the time and the items that differed never did so by more than 10%. These results indicate that the Tinetti Assessment Tool has good interrater reliability.

### **VALIDITY**

The Tinetti POMA test has been determined to be a valid test in elderly populations amongst other populations and those with mild to moderate dementia.

### REFERENCES

Lewis C. Balance, Gait Test Proves Simple Yet Useful. P.T. Bulletin, 1993; 2/10:9 & 40 Tinetti ME. Performance-oriented Assessment of Mobility Problems in Elderly Patients. J Am Geriatr Soc 1986; 34:119-126.

Tinetti ME, Williams TF, Mayewski R, Fall Risk Index for elderly patients based on number of chronic disabilities. Am J Med 1986:80:429-434

Cipriany-Dacko LM, Innerst D, Johannsen J. Interrater reliability of tinetty balance scores in novice and experienced physical therapy clinicians. Arch Phys Med Rehabil. 1997; 78(10): 1160-1164

Tooper AK, Maki BE, Holliday PJ. Are activity-based assessments of balance and gait in the elderly predictive of risk of falls and/or type of fall? J Am Geriatr Soc 1993; 41: 479-487

Kegelmeyer DA, Kloos AD, Thomas KM, Kostyk SK. Reliability and validity of the tinettu mobility test of individuals with Parkinson Disease. Phys Ther 2007: 87(10): 1369-1378.

| Participant Number: | Date: | <br> |
|---------------------|------------|------|
| | Evaluator: | |

### POMA BALANCE SECTION

Resident is seated in hard, armless chair;

| TASK | DESCRIPTION | SCORE (0-2) |
|---|---|---|
| 1 CITTING DALANGE | Leans or slides in chair | |
| 1. SITTING BALANCE | Steady, safe | |
| | Unable without help | |
| 2. RISES FROM CHAIR | Able, uses arms to help up | |
| | Able without using arms | |
| A AFFEN (PEG TO PIGE | Unable without help | |
| 3. ATTEMPTS TO RISE FROM CHAIR | Able, requires > 1 attempt | |
| TROW CHAIR | Able to rise in 1 attempt | |
| 4. IMMEDIATE | Unsteady (swaggers, moves feet, trunk sways) | |
| STANDING BALANCE | Steady but uses walker or other support | |
| (first 5 seconds) | Steady without walker or other support | |
| | Unsteady | |
| 5. STANDING | Steady but wide stance (heels 4 inches apart) | |
| BALANCE | and uses cane or other support Narrows stance without support | |
| 6. NUDGED (subject | | |
| at max position with | Begins to fall | |
| feet as close together | Staggers, grabs, catches self | |
| as possible, examiner pushes lightly on subject's sternum with palm of hand 3 times) | Steady | |
| 7. EYES CLOSED (at | Unsteady | |
| max position – see #6) | Steady | |
| | Discontinuous steps | |
| 8. TURNING 360 | Continuous steps | |
| DEGREES | Unsteady (grabs, swaggers) | |
| | Steady | |
| | Unsafe (misjudged distance, falls into chair) | |
| 9. SITTING DOWN | Uses arms or not a smooth motion | |
| | Safe, smooth motion | |
| | <b>Total Balance Score</b> | |

### **POMA GAIT SECTION**

Initial Instructions: Subject stands with examiner, walks down the hallway or across the room, first at "usual" pace, then back at "rapid but safe" pace. Use usual walking aid.

| TASK | DESCRIPTION | SCORE (0-2) |
|---|---|---|
| 10. INITIATION | Any hesitancy or multiple attempts to start | |
| GAIT (immediately after told to "go) | No hesitancy | |
| - | RIGHT swing food does not pass left stance foot with step | |
| | RIGHT foot passes left stance foot | |
| | RIGHT foot does not clear floor completely with step | |
| 11. STEP LENGTH | RIGHT foot completely clears floor | |
| AND HEIGHT | LEFT swing foot does not pass right stance foot with step | |
| | LEFT foot passes right stance foot | |
| | LEFT foot does not clear floor completely with step | |
| | LEFT foot completely clears floor | |
| 12. STEP | RIGHT AND LEFT step length not equal-estimate. | |
| SYMMETRY | RIGHT AND LEFT step appear equal | |
| 13. STEP | Stopping or discontinuity between steps | |
| CONTINUITY | Steps appear to continue | |
| 14. PATH (estimated | Marked deviation | |
| in relation to floor tiles, | Mild/moderate deviation or uses walking aid | |
| 12-inch diameter. Observe excursion of 1 foot over about 10 feet of the course) | Straight without walking aid | |
| | Marked sway or uses walking aid | |
| | No sway – but flexion of knees or back, | |
| 15. TRUNK | or spreads arms out while walking | |
| | No sway, no flexion, no use of arms, | |
| | and no use of walking aid | |
| 16. WALKING STANCE | Heels apart | |
| 10. WALKING STANCE | Heels almost touching while walking | |
| | <b>Total Gait Score</b> | |

### **POMA SORING SECTION**

| Score – Balance | /16 |
|-----------------|-----|
| Score – Gait | /12 |
| Score – Total | /28 |

| Assessor Signature & Title: |
|-------------------------------|
| Location During Assessment: _ |

### **Risk Indicators:**

≤18 High

19-23 Moderate

≥24 Low

### 17.1.3: Two Minute Walk Test (TMWT)

### Two Minute Walk Test

### **General Information:**

- ✓ Individual walks without assistance for 2 minutes and the distance is measured from the start of timing when the individual is instructed to "Go"
- ✓ Stop timing at <u>exactly 2</u> minutes
- ✓ Assistive devices can be used but should be kept consistent and documented from test to test
  - o If physical assistance is required to walk, this **should not be** performed
- ✓ A measuring wheel is helpful to determine distance walked should be performed at the fastest speed possible

### **Set-up and equipment:**

- ✓ A measuring wheel is helpful to determine distance walked should be performed at the fastest speed possible
- ✓ Ensure the hallway free of obstacles
- ✓ Functioning stopwatch ready.

### **Participant Instructions**

"Cover as much ground as possible over 2 minutes. Walk continuously if possible, but do not be concerned if you need to slow down or stop to rest. The goal is to feel at the end of the test that more ground could not have been covered in the two minutes."

Minimal Detectable Change (MDC) – 12.2m (90% Confidence)<sup>1</sup> Normative Data (LTC) – 77.5m (±25.6)

### Two Minute Walk Test (TMWT)

| Participant Number: | | Date: | |
|---|---|---|---|
| | Evalua | tor: | |
| | eed to slow down o | e over 2 minutes. Walk continuously or stop to rest. The goal is to feel at to the two minutes to the two minutes. | the end of the test that more |
| Distance Walked: _ | | (metres) | |
| Gait Aid Used? | YES | NO | |
| If yes, what was u | sed: | | |
| Notes: | | | |
| Assessor Signatur | e & Title: | | |
| Location During A | l cceccment: | | |

### 17.1.4: Knee Range of Motion (ROM)

### **Knee Range of Motion Test (ROM)**

**Description:** Assess the range of motion of the patient's knees.

**Equipment:** Examination bed, goniometer, rolled towel

### **Therapist Instructions:**

### **Knee Extension:**

-Have the patients placed in supine position, hips at neutral and with the knee in extension

-A rolled towel is placed under the calcaneus to maximize knee extension

-The goniometer's fulcrum is centered over the lateral condyle of the femur. The arms are aligned with the greater trochanter and lateral malleolus.

-The angle formed by these landmarks was the maximal angle of extension

### **Knee Flexion:**

-The patient lifts their leg off of the towel and places their foot flat on the examination table. The patient brings their foot as close as possible toward their hip closing the angle of their knee as much as possible.

- The goniometer's fulcrum is centered over the lateral condyle of the femur. The arms are aligned with the greater trochanter and lateral malleolus.

-The angle formed by these landmarks was the maximal angle of flexion

-The patient might need assistance, aid as necessary

### **Resident Instructions:**

-Please lie on this bed and place your ankle on this towel and extend your knee as much as possible

-I'm just going to find a portion of your hip

-Now, if you could bend your knee, bring your foot as close as you

can to your hip and keep your foot flat on the table.

### References

Norkin CC, White DJ. Measurement of Joint Motion: A Guide to Goniometry. 3<sup>rd</sup> ed. Philadelphia: FA Davis Company; 2003.

### **Knee Range of Motion (ROM)**

| Participant Number: | Date: | |
|----------------------------------------------------|-------|---|
| Evaluator: _ | | |
| Max extension left knee: | | |
| Max flexion left knee: | | |
| Max extension right knee: Max flexion right knee: | | |
| Assessor Signature & Title: | | |
| Location During Assessment: | | _ |

### **Appendix B:** Participation Outcomes

### 17.2.1: BikeAround Session Evaluation

### **Bike Around Session Evaluation**

| <b>Participant Number:</b> |
|----------------------------|



| Date | Baseline<br>Mood (#) | Baseline<br>Time | Follow Up<br>Mood (#) | Follow<br>Up Time | Distance<br>Travelled (KM) | Pedometer<br>Time | Who Facilitated? |
|---|---|---|---|---|---|---|---|

2

Level of resistance (please circle)  $\rightarrow 0$ 

1

3

Ļ

6

5

7

8

| | | 10 | 20 | 30 |
|---|---|---|---|---|
| | Interest in others (staff, cycle hosts, etc.) | | | |
| Interest | Without prompts offers support of a peer | | | |
| Interest | Acknowledges support from a peer | | | |
| | While engaged sustains attention | | | |
| Attention | Requires verbal prompting or cueing | | | |
| Attention | Initiates or engages in conversation | | | |
| Pleasure | Relaxed body language, smiles, and laughs | | | |
| Pleasure | Verbalizes sense of pleasure | | | |
| | Anger | | | |
| Negative Affect | Physical signs of agitation | | | |
| Negative Affect | Verbalizes feeling anxious | | | |
| Sadness | Behavioral signs of sadness | | | |
| Sauness | Verbalizes feeling sad | | | |
| | Non-verbal expression of pride | | | |
| Self Esteem | Verbal expression of satisfaction | | | |
| Sell Esteelli | Inferred prideful reminiscence | | | |
| | Verbal expression of normalcy | | | |
| Normaley | Non-verbal expression of social normalcy | | | |
| Normalcy | When joining or leaving, interacts with others | | | |

4- Always

3- Most of the time

2- Some of the time

1- Rarely

0 – Never

Resident expresses an interest to continue with program What seating adjustments were made for the resident?

Yes

No

What location did the resident visit?

### **Resident Refusal Form**

Please mark Resident on this list if they were;

- (A) Absent from participation

(i.e. Out with family, in another program, in shower, etc.)

OR

- (C) Chose to not participate on a day when they were scheduled

(i.e. They verbally told you they didn't want to participate)

OR

- (SL) Sleeping

(i.e. Unable to wake up or too drowsy)

OR

- (S) Sick

(i.e. they were not feeling well, or a nursing staff mentioned they were not feeling well)

| Date | Time of Day | Participant<br>Number | Resident Reason | Volunteer<br>Name |
|---|---|---|---|---|
| June 1st | 11:00am | PN22 | (C)<br>Didn't want to come | Becky |

EX.

### **Appendix C:** Field Notes - Qualitative Outcome

| Participant ID: | |
|---|---|
| Date: | Time: |
| <b>Observations:</b> (If completing these forms during a like discussions that participants are having with a changes in behaviour or mood; location selection, at the start of a session if field notes can be taken.) | others, including research staff or other staff;<br>if applicable; and so on. Always ask participants |
| The location the participant went: | |
| Did the participant pick this location (Circle): | Yes No |
| Was there a change in the participant's mood | (Circle): Yes No |
| Please Describe this change: | |
| Other observations: | |

### **Appendix D:** Medical Chart Data Outcome Extraction Sheet

| rticipant Number: | Date: | |
|---|---|---|
| Chart Reviewer: | | |
| level of consciousness, and exec | ance Scale (CPS) combines infort<br>cutive function, with scores rang<br>as been shown to be highly corre | ing from 0 (intact) to 6 (very |
| Journal of Gerontology: Medical Scie | | - |
| <u>SCORE</u> | <b>Date Evaluated</b> | <u>Notes</u> |
| Revised Index of Social Engagen | ment (RISE) | |
| on being at ease interacting wit<br>invitations, pursuing involveme<br>to interactions. Scale scores ran | cial Engagement (RISE) is a med<br>th others, being at ease doing pla<br>ent in life of facility, initiating into<br>the from 0-6 with higher scores is<br>cility. The index is a revised yers | inned activities, accepting<br>eractions and reacting positive<br>indicative of greater social |
| | veloped for an earlier version of t | ion of the Index of Social<br>the RAI for long term care |
| Engagement (ISE) that was dev | | |
| Engagement (ISE) that was dev facilities. | reloped for an earlier version of t | the RAI for long term care |
| Engagement (ISE) that was dev facilities. | reloped for an earlier version of t | the RAI for long term care |
| Engagement (ISE) that was dev facilities. | reloped for an earlier version of t | the RAI for long term care |

BikeAround Study Protocol – Version 8.0, May 2019

| Participant Number: | Date: |
|---|---|
| Chart Reviewer: | |
| Current Medication list: Compile a list of all of the medications each particle. | articipant is on (both amount and frequency) |
| Medication Name | <b>Dosage information</b> |
| Medication Name | Dosage information |
| Medication Name | Dosage information |

### **Activity Pro Data**

### **Extraction Sheet**



| <u>Participant Numb</u> | er: | |
|---------------------------|--------------------|-------|
| <b>Project Phase:</b> | | |
| <b>Date Range:</b> | | |
| Overall Engageme | ent Score: | |
| Self-Directed Scor | <u>·e:</u> | |
| <b>Total Minutes of I</b> | Engagement: | |
| Number of Activit | ty Participations: | |
| Category | Total Number | Notes |
| C (Chose not to attend) | | |
| S (Sick) | | |
| SL (Sleeping) | | |
| A (Absent) | | |
| Data Fytra | | |
| Data Extra | acted By: | |

### **Appendix E**: Cross-Over Study Design Diagram



### **Appendix F:** Newsletter Paragraph

The Glebe Centre, in partnership with the University of Ottawa and Bruyère Research Institute, is excited to begin recruitment for a research project that will provide residents with an opportunity to engage in a cycling (stationary) activity that is combined with a virtual trip to anywhere Google Maps have been...anywhere around the world. These virtual images may help engage and immerse residents into the activity. We are looking to observe how residents engage in this activity and whether it can improve their balance and mobility. Whether your resident has participated in this activity before or not, feel free to contact Susan Zorz at <a href="mailto:SZorz@glebecentre.ca">SZorz@glebecentre.ca</a> or 613.238.2727 X 323 for more information.

### **Appendix G:** Recruitment Script for Staff

### When discussing with the resident:

### LTC Staff:

"I would like to let you know that there is a research project underway here at The Glebe Centre that you may be eligible for. Your decision to hear more about this project will not impact the care you receive here at The Glebe Centre. It is completely voluntary, and you have the right to stop participation at any time. Would you like to hear more about this research project?"

If YES:

"Wonderful, thank you! Can I have your verbal consent to pass your information to a member of the research team? They will come by to see you in a few days to provide you more information about this project."

### If NO:

"No problem at all. Again, this does not impact the care that you receive here at The Glebe Centre."

### If questions arise regarding this project:

"As I am not directly involved with this research project, I would have to defer you to the research team to have your questions answered."

### When calling the SDM:

\*\*After confirming you are talking to the SDM for the resident:

| LTC Staff | • | |
|---|---|---|
| "I would la | ike to let you know that there is | a research project underway at The Glebe Centre |
| that | <u>(insert name here)</u> | is in. Your decision to hear more about this |
| project wil | ll not impact the care they recei | ive here at The Glebe Centre. It is completely voluntary |
| and they h | ave the right to stop participati | on at any time. Would you like to hear more about this |
| research p | roject?" | |
| If YES: | | |
| "Wonderfi | ul, thank you! Can I have your | verbal consent to pass your contact information to a |
| member of | the research team? They will c | contact you in a few days to provide you more |

member of the research team? They will contact you in a few days to provide you more information about this project."

If NO:

"No problem at all. Again, this does not impact the care that <u>(insert name here)</u> receives here at The Glebe Centre."

### If questions arise regarding this project:

"As I am not directly involved with this research project, I would have to defer you to the research team to have your questions answered."

### When emailing the SDM

\*\*After confirming you are using the email on file for the SDM:

| LTC Staff: |
|---|
| Hello(Insert name of SDM), |
| "I would like to let you know that there is a research project underway at The Glebe Centre that <u>(insert first name here of resident)</u> is in. Your decision to hear more about this project will not impact the care they receive here at The Glebe Centre. It is completely voluntary, and they have the right to stop participation at any time. If you would like to hear more about this research project please reply to this email and a member of the research team will contact you in a few days to provide more information. |
| Sincerely, |
| (insert your name) |
| If YES reply: "Wonderful, thank you! They will contact you in a few days to provide you more information about this project." If NO reply: |
| "No problem at all. Again, this does not impact the care that (insert name |
| <u>here)</u> receives here at The Glebe Centre." If questions arise regarding this project: |
| "As I am not directly involved with this research project, I would have to defer you to the research team to have your questions answered." |

### **Appendix H:** Recruitment Script for RA

| 1. Introduction of Research Te | eam Member to SDM/POA: | |
|---|---|---|
| "Good morning/ Good afternoon/ Go | ood evening Mrs./Mr./Ms | . <i>My</i> |
| name is | I'm one of the research | ers for an activity study |
| happening at The Glebe Centi | re that | mentioned to you, and |
| indicated to me that your love | d one might be interested in p | participating". |

### 2. Introducing the Study

"This study involves your loved one using a stationary bike while supervised during their daily activities. This bike is safe and effective for encouraging increased activity for older adults. This is not a real exercise bike, but rather a modified version that your loved one will sit on his own chair and use their arms and legs to engage in activity. This study will go for 18 weeks. Your loved one will either have the opportunity to use this bike for the first 6 weeks or delayed to the second group during the last 6 weeks. Whichever group they are randomized to, they will have the opportunity to participate. During these sessions, your loved one will be helped to the bike by myself, a volunteer, a recreation therapist or a staff member on the unit. Their participation is optional every day. During their pedalling, they will be immersed into a large dome that can display images captured on Google Street View. They can select where in the world they would like to pedal with help from the cycle host. If you decided to allow your loved one to participate, we would love to have your help to create a list of fun places for them to visit. Our hope is that residents who participate in this program will experience overall improvements in their quality of life."

### 3. Consent

"Would you be interested in having your loved one participate in this project?" (If yes, proceed to #4 If no, proceed to #5a).

### 4. Follow-Up for Written or Oral Informed Consent

- "When might be the next time you'll be visiting The Glebe Centre, in order for one of the researchers to meet with you to read and sign the full Informed Consent form?

  Alternatively, we can record your oral consent for your loved one to participate and send you the form electronically for your information."
- \*(Also give option to send form electronically first, and then follow-up with another phone call for oral consent if the SDM/POA prefers).
- \*\*Note, the researcher will also have the Informed Consent form nearby in order to answer any other questions directly from the information provided in the form \*\*\*

### 5. Finish the call

- a. "No problem at all! This decision does not impact the care your loved one will receive here at the Glebe Centre. Once the project is completed, your loved one will still have the option of using the bike, without being part of any research project."
- b. "Thank you very much for your time."

### **Appendix I:** Participant Consent Form

The following document will be used solely with residents that have the ability to provide informed consent. This will be decided by the health care team.



Participant Consent Form May2019\_Clea

### **Appendix J: SDM Consent Form**

The following document will be used with substitute decision makers for residents that do not have the ability to provide informed consent. This individual must be identified in the resident's file as a substitute decision maker.



### **Appendix K:** Master Code List

\*This mater code list will be password protected and only saved on the secure server at The Glebe Centre.

| Resident Name | Participant<br>Code | Room Number | SDM | SDM Contact<br>Number |
|---|---|---|---|---|
| Jennie Smith | PN01 | 424 | Johnnie Smith | 613-555-5555 |

### **Appendix L:** CABHI Budget

| Project End: |
|------------------|
| 2019-08-31 |
| Institution |
| The Glebe Center |

Funding from CABHI
The maximum funding available for projects selected in this call for innovations is \$50,000 (CAD). The SPARK Program will be funding projects that are scheduled to run for 6 to 12 months, starting in February 2018. CABHI funding will be attached to project milestones and deliverables. Funding will flow to the applicant's host organization. The host organization will be accountable for the applicant's completion of project milestones and deliverables as well as performance

### In-Kind Contributions

Funding from the Host Institution

CABHI releases an initial payment of 90 per cent of its funding at the start of the project. A holdback of 10 per cent will be released upon project completion and receipt of final progress and financial reports, outcomes and attestation from the host organization regarding the use of funds.

# No specific amount of matching funds from the Host Institution is required to apply for the program. The Host Institution may contribute in cash or in-kind, either from its own sources or through other funding sources. For example, applicants might show evidence of government, industry partner or institutional commitment through a blend of cash and/or in-kind contributions such as office space, equipment, connectvity, staff salaries, etc.

quested from CABHI (SCAD, should match amount indicated in application)
cured from other sources (in-kind, valued in SCAD)\*(Specify clearly the sources of all in-kind contributions; add and/or delete rows as needed)
Program Facilitator - 18 hours/week salary plus employer related costs 49,754.00 26,019.23 2,400.00 7,867.34

| Program A | Project Lea | Salaries and b | Program F | Salaries and b | a) Personnel | Important: A<br>Sample tab f | Commentary<br>"http://www | EXTIMATED |
|---|---|---|---|---|---|---|---|---|
| Program Assistant @16/hour x 22.5 hours/week for 52 weeks + 21.5% employer related costs | Project Lead (19.00/hour x 22.5 hours / week for 52 weeks + 21.5% employer related fees) | Salaries and benefits (new personnel) | Program Facilitator (18 hours/week @ 22.88/hour x 52 weeks + 21.5% employer related costs) | Salaries and benefits (existing personnel) | | Important: All expense categories (e.g., Materials and Supplies) need to be itemized. For example, an expense entry within "Materials & Supplies" would require the name of the material/supply, quantity and price per quantity. See Sample tab for further information. | Commentary: Eligible costs are expenses that are directly related to the project, are incurred at or on behalf of the Host Institution, and achieve its milestones and deliverables, subject to the limitations set out in the "http://www.ccabhi.com/wp-content/uploads/Spark-Program-Eligible-Expenses-Guideline.pdf". Funding will flow to the applicant's host organization. | EXTIMATED PROJECT EXPENDITURES |
| \$ 22,744.80 | \$ 27,009.45 | | \$ 26,019.23 | | | ıls & Supplies" would r | and achieve its milesto<br>plicant's host organiza | AMOUNT<br>(\$CAD) |
| CABHI | CABHI | | The Glebe Centre | | | equire the name of the m | nes and deliverables, subtion. | Source Name (if more<br>than one, breakdown<br>by %) |
| | | | \$ 26,019.23 | | | aterial/supply, quantity an | ject to the limitations set o | In-kind Contributions (If applicable, see note in "Requested/Secured Funds") |
| \$ 22,744.80 | \$ 27,009.45 | | | | | d price per quantity. See | ut in the | Cash |

| \$ 49,754.25 | \$ 36,786.57 | | \$ 86,540.82 | GRAND TOTALS |
|---|---|---|---|---|
| | | | | Total other costs |
| | | | | e) Other |
| | | | \$ . | Total travel costs (pre-approved by GABH) |
| | | | | International travel |
| | | | | Travel within Canada |
| | | | | d) Travel |
| | | | \$ | Total equipment costs |
| | | | | c) Equipment |
| \$ | \$ 10,767.34 \$ | | \$ 10,767.34 | Total non-personnel related costs |
| | | | | Other expenditures (provide detail) |
| | | | | Minor equipment |
| | | | | Meetings and events |
| | 3 /,00/,34 | THE GIEDE CEHTE | 3 /,86/.34 | autiun resources, rinances and musing support (10% of acts profess cost) |
| | | $\perp$ | | Office and administrative |
| | | | | Participant costs |
| | | | | Professional and technical services |
| | \$ 2,400.00 | The Glebe Centre | \$ 2,400.00 | Camino Support - The Glebe Centre pays a monthly maintenance fee to Camino for the Bikeskround, this cost will continued to be |
| | | | | Hardware, software and IT support |
| | | | | Site preparation and training |
| | \$ 500.00 | The Glebe Centre | \$ 500.00 | Paper, photocopier, printers, communiques |
| | | | | Materials and supplies |
| | | | | b) Non-Personnel Related Costs |
| \$ 49,754.25 | \$ 26,019.23 \$ | | \$ 75,773.48 | Total personnel costs |
| | | | | Other expenditures (provide detail) |

### Appendix M: Summary of Fall Prevention Program at The Glebe Centre

This program focuses on reducing the incidence of residents' falls and mitigating risks of falls through a resident focused, team approach which ensures that a resident's environment and social, physical, cognitive and emotional strengths are supported. The program ensures team training, communication and effective care planning. This is an interdisciplinary program involving nursing and program staff, physician/pharmacist, dietician, physiotherapist, housekeeping staff and the resident/POA. They communicate regarding their planned interventions and evaluation of resident progress and outcomes in falls prevention through documentation. This program works in collaboration with the Centre's Restraint reduction and Restorative care programs.

Every Resident's Fall Risk is assessed using Scott Fall Risk Assessment by registered nursing staff on admission, after a fall and when there is a significant change in condition. Based on the assessment residents are categorized into High and Very High risk and Interventions are targeted in areas contributing to falls.

A number of fall prevention tools are used in the facility such as motion sensors, seat belt alarms, bed sensor pads. Hourly rounding of residents to prevent falls and avoid use of restraints is also part of the daily routine. Equipment such as fall mats, hip protectors, low electric bed are also used to prevent significant injury in case of a fall.

The Restorative Program also works along with the Fall Prevention Program in identifying those at high risk for falls and exercises are carried out by nursing staff seven days a week to strengthen lower extremities and prevent falls. Along with Nursing, Physiotherapy staff and program facilitators are also involved in providing balance and strength exercises which area core component of the Fall Prevention Program to reduce the number of falls. Residents' Fall Risk is communicated at the Interdisciplinary Care Conferences to keep families (POA/ADM) informed of the actions taken to prevent falls.

The Nurse Practitioner assigned to The Glebe Centre is referred to one-time fallers to rule out medical causes to prevent further fall. The Co-coordinator of Nursing Program audits all falls on a daily basis and acts as a resource to the rest of the staff in identifying risk areas, suggesting new interventions and also responsible for reviewing the program on an annual basis.

### Appendix N: Poster for presentation in main fover

Poster was presented at 2018 Regional Geriatric Annual General meeting and will be used to promote study by being placed in main foyer of The Glebe Centre to advertise the research.



The Globe Control was founded in 1868 as 0 hairb's first home for the Agod and 2018 marks our 132nd arrive sary of dedication to seniors through the provision of services, tability-based care and personal support.

## The Glebe Centre

Susan Zorz, Director of Resident Services and The Glebe Centre Team

Residents in Long Term Care Using the Jdome BikeAround to Impact Health and Wellness for

## Our main goal for this project is to assues the differentiates of participation in the BioArcurd program as a viote owner so intervention that will improve functional ability and measure significant positive changes with mobility assues and quality of intervention that will improve functional ability and measure significant positive changes with mobility assues and quality of The main goal for funding this project is to support a project lead and program assistant to ensure that we can develop this program formal exercise physiology in execution program which can be implemented in our forme and a revention

# CABHI: Spark Grant Winners!



Past dens two excross regularly lose less polit monde energy and microsoft function resulting in realisce resk of "a lis. Qualitative, yerd in distriety we see the positive result that in Yadeneen; in this program has all easy has on the artistycers. Our resultarph to partify you'd new televe in the tine.

# Features of the BikeAround

One of the biggest challenges in health care is to offer meaningful activities.



The Rissak word has a personneter attached to 1 so see aberate to add another element of excitement of the program by tracking how for participants are traveling during cash session.

# **Current Stages of Development**

Front including contained to assess mod by and apply universal rails prevention problems a approximate. We believe that the additional intervention of the Diselecting program to our current talk management program an important impact on reducing the number of talk in our home.

## **Supporting Evidence**

An exercise program structor include the basic comparants of physical fluxes, from muscle strength and floatility to be since, coordination and stamma. Worth Lagdeneim Helbostadt

A resortier will be retailed and under die der best auch its intell behand Assessment bed and the Scott all Black Assessment Jobb Way will also measure at retailenses of the Billed round by monitoring the CIT countriefy reports and our Bit Aufüg reporting mechanismes. Additionations are not induced monopolitic for interesant sees and appoints result and mentionations, more independence and cast by in activities of they before Using Blackround technology we will explane the impact on fail reduction for excipt with a griff auth exquitive assessment of set cheen a health conditions.

**Key Outcomes** 

A program protect , assessment foot and exclusion have been developed. We also use the Wong Baker Scale to evaluate Resident Satistication. consistion, that in gradients who have directly concessing thorasters. Come has no measure include. This is the best day every." I distribute I would see go beats," I sharks so much for this, I am neally gratefull and "This was familiation." One resident was singing and telling dionles all the way book to the unit.

BikeAround at the Glebe Centre